CLINICAL TRIAL: NCT02429167
Title: Double Blind, Randomized, Sham Controlled Study of Safety and Effectiveness of the Portable Neuromodulation Stimulator (PoNS) Device for Cranial Nerve Noninvasive Neuromodulation Training for Chronic Balance Deficit Due to Mild/Moderate TBI
Brief Title: Study of Safety and Effectiveness of PoNS Device to Treat Chronic Balance Deficit Due to Traumatic Brain Injury (TBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helius Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NHC-TBI-PoNS-RT001
Record Dates: First submitted 2015-04-20; First posted 2015-04-29 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Traumatic Brain Injury; Chronic Balance Disorder
Keywords: Traumatic Brain Injury; Neuromodulation; Chronic Balance Disorder
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PoNS Device (Experimental): Cranial nerve non-invasive neuromodulation via PoNS device. The system delivers 19 V pulses to the tongue (a nominal 5.5 kilo-ohm load).
  Interventions: Device: Cranial nerve non-invasive neuromodulation via PoNS device
- Sham PoNS Device (Sham Comparator): The sham control device appears physically identical but uses a modified stimulus waveform parameter set designed to elicit a mild tactile sensation while minimizing the net energy delivered, thereby providing minimal, if any, cranial nerve non-invasive neuromodulation via PoNS device
  Interventions: Device: Sham PoNS device

INTERVENTIONS:
Device: Cranial nerve non-invasive neuromodulation via PoNS device — The PoNS is a medical device worn around the neck. The controller contains the pulse generator and a user interface. The mouthpiece, held to the top of the tongue, contains 143 circular gold electrodes that deliver a mild, controlled electric stimulation to the subject. While the subject is receiving stimulation, they will perform increasingly difficult balance, posture, gait, and movement control tasks designed to challenge existing abilities. Each training session takes approximately one hour to complete, and is separated by an interval of 2-2.5 hours.
  Arms: PoNS Device
Device: Sham PoNS device — The PoNS is a medical device worn around the neck. The controller contains the pulse generator and a user interface. The mouthpiece, held to the top of the tongue, contains 143 circular gold electrodes that deliver a mild, controlled electric stimulation to the subject. The sham control device is physically identical but uses a modified stimulus waveform parameter set designed to elicit a mild tactile sensation while minimizing the net energy delivered, minimizing any neuromodulatory effect. While the subject is receiving stimulation, they will perform increasingly difficult balance, posture, gait, and movement control tasks designed to challenge existing abilities. Each training session takes approximately one hour to complete, and is separated by an interval of 2-2.5 hours.
  Arms: Sham PoNS Device

SUMMARY:
The purpose of this study is to determine if clinic and home training with a study device will improve a balance deficit. The study device is called Portable Neuromodulation Stimulator (PoNS). The study device will be placed on the tongue to deliver nerve stimulation. The study is testing if use of the study device in conjunction with physical therapy will improve balance and gait in patients suffering from a TBI. The effects of using the device and undergoing therapy will be measured using standardized tests of movement control, gait, headache and other TBI symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-65 years of age
* Documentation on initial TBI (defined as closed-head, non-penetrating, blunt, whiplash, or explosive blast-induced brain injury) severity (at time of injury): Glasgow Coma Scale (GCS) score 9-15, with loss of consciousness < 24 hours, post-traumatic amnesia ≤7 days, or hospital admission ≤ 7 days post TBI
* If female, subject is not pregnant, not lactating, has a negative pregnancy test prior to receipt of the PoNS™ device, and agrees to use contraception from screening to end of the study
* Balance disorder with SOT composite score at least 16 points below normal resulting from a mild/moderate TBI without any concomitant pathologies
* At least 1 year post injury
* Stable neurologic status
* Prior participation in a focused physical rehabilitation program for TBI and deemed by their treating clinician/themselves to have reached a plateau
* Able to walk continuously on a treadmill for 20 minutes, level grade and at any speed, with support if needed
* Access to a treadmill and commitment to utilize this for the at-home portion of the study
* Able to understand the study procedures and give informed consent
* Willing and able to adhere to the study schedule
* Willing to complete a neuropsychological evaluation prior to inclusion

Exclusion Criteria:

* Medical finding from screening history and physical examination that is clinically significant or would otherwise impact patient safety or data integrity
* Medical finding from prior neuroradiologic study or recent MRI that is significant or that would impact patient safety or data integrity
* Planned use or use of any investigational product, pharmaceutical or device within 30 days preceding receipt of the PoNS device and during the entire study
* Balance or gait deficits due to lower extremity injury or neurological condition other than TBI
* Penetrating brain injury, craniotomy or refractory subdural hematoma
* Oral health problems at the time of recruitment
* Oral surgery within 3 months of screening
* History of oral cancer
* Non-removable metal orthodontic devices that could interfere with PoNS use
* Presence of metallic implant or other MRI-incompatible device
* Blood pressure abnormalities considered clinically significant
* Use of Coumadin or other anticoagulant except aspirin in the last 6 months
* Untreated or undiagnosed diabetes
* Diabetic neuropathy
* Active or recent (within 1 year) treatment for any cancer, excluding basal cell carcinoma.
* Neurological disorders other than those attributed to the primary diagnosis (neurodegenerative diseases such as Multiple Sclerosis, Parkinson's disease, Alzheimer's disease or other dementia, Amyotrophic Lateral Sclerosis)
* History of epileptic or other seizure disorders
* Known ischemic heart disease and/or history or atrial or ventricular arrhythmias with or without syncope
* Any other untreated or unstable acute or chronic, clinically significant medical condition for which the subject is currently undergoing treatment that the study investigator deems unsuitable for inclusion
* Use of a lower extremity biomechanical prosthetic with the exception of a splint for foot drop
* Females who are pregnant, lactating, or planning to become pregnant during the study
* Chronic use of any potentially interfering medication, or use of any medication that would compromise the ability to function or perform the study activities
* Addition of and/or major change in type or dosage of any prescription medication within 3 months prior to receipt of the PoNS device
* Active alcoholism. The study investigator will have the right to exclude subject participation if the subject seems intoxicated at time of screening and/or during any study appointment.
* History of drug abuse will be assessed
* Recent history of smokeless tobacco use
* Any reason that may be a threat to health or safety
* Any finding in the neuropsychological evaluation that makes the subject unsuitable for inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Response to treatment defined as an 8 point change in the Sensory Organization Test (SOT) from baseline | 5 weeks after the start of the intervention
  The SOT is an objective, automated measure of sensory-motor integration that evaluates the functional contribution of the somatosensory, visual, and vestibular components of balance. A composite score is calculated and compared with a database normalized for age and height.

SECONDARY OUTCOMES:
Increase in SOT score from pre-training SOT score at the end of 2 weeks in lab training | Two weeks after start of the intervention

OTHER OUTCOMES:
Frequency of falls | Daily for 5 weeks
Frequency of headaches | 5 weeks
  Frequency of headaches will be assessed using the headache disability index

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Orlando Health, Orlando, Florida
  - Oregon Health and Science University Center for Regenerative Medicine, Portland, Oregon
- The Montreal Neurofeedback Center, Montreal, Quebec, Canada